CLINICAL TRIAL: NCT01263769
Title: A Phase II Clinical Trial Examining the Impact Of Neoadjuvant Axitinib On Primary Tumor Response In Patients With Locally Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Neoadjuvant Axitinib in Locally Advanced Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0072; NCI-2011-00279 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Kidney Cancer
Keywords: Locally advanced clear cell renal cell carcinoma; AG-013736; Axitinib; Radical nephrectomy
MeSH Terms: conditions — Kidney Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axitinib (Experimental): Axitinib Starting dose: 5 mg by mouth twice each day for 12 weeks.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Starting dose: 5 mg by mouth twice each day for 12 weeks.
  Other Names: AG-013736

SUMMARY:
The goal of this clinical research study is to learn if axitinib can help to control kidney cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Axitinib is designed to decrease blood supply to the tumor, which may slow tumor growth.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take axitinib by mouth 2 times a day every day for 12 weeks. The dose may be changed based on any side effects you may have. You should take the drug about 12 hours apart. You should take the pills at about the same time each day. If you vomit anytime after taking a dose, you must not "make it up" with an extra dose, but instead take the next dose as previously scheduled. Any missed dose may be taken late up to 3 hours before the next scheduled dose, otherwise, it should be skipped.

A blood pressure monitor will be given to each participant for home use. You will be given instructions and shown how to monitor your blood pressure.

You will be provided with a calendar to record the date and time of each dose, and your blood pressure reading before taking the drug. Missed doses should also be recorded. You must also bring the study drug bottle to each study visit so the research nurse can count any remaining pills.

A drug list will be given to you to record drugs taken within 4 weeks before you enrolled on the study and while on study. A new list will be provided during each clinic visit. You should not start a new prescription or over-the-counter drug before talking with the study doctor, except in the case of a medical emergency.

Study Visits:

At Week 1:

* You will be asked about any drugs you may be taking.
* Your performance status will be recorded.
* You will complete the questionnaire about kidney cancer care. This questionnaire will take about 5 minutes to complete.
* Women who are able to become pregnant will have a blood (about 1 teaspoon) or urine pregnancy test.

At Week 3:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status will be recorded.
* You will have an ECG.
* Blood (about 2 tablespoons) will be drawn for routine testing to check your thyroid function.
* Urine (about 2 tablespoons) will be collected for routine testing.
* You will complete the questionnaire about kidney cancer care.

At Weeks 5 and 9, you will be called and asked if you have had any side effects. This call should take about 10 minutes.

At Weeks 7 and 12:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine testing and to check your thyroid function.
* Urine (about 2 tablespoons) will be collected for routine testing.
* You will complete the questionnaire about kidney cancer care.
* You will have a CT scan of chest and abdomen to check the status of the disease.
* At Week 12 only, you will have an ECG.

At Week 13, you will have surgery to remove the kidney tumor. You will receive a separate consent form for this surgery.

At Week 19:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine testing and to check your thyroid function.
* You will complete the questionnaire about kidney cancer care.
* You will have a CT scan of chest and abdomen to check the status of the disease.
* If you have been treated for high blood pressure while taking the drug, your blood pressure will be monitored and your blood pressure medication will be reduced. Once your blood pressure reaches a certain level, this will be managed by your primary care doctor.

After Week 19, every 4 months (+/- 2 weeks) for the first 1 year, every 6 months (+/- 2 weeks) for the third and fourth year, then every year (+/- 1 month) for a total of 5 years post surgery:

* Your medical history will be recorded.
* You will have a physical exam.
* Your performance status will be recorded.
* You will have a CT scan of the chest and abdomen to check the status of the disease.
* Blood (about 2 tablespoons) will be drawn for routine testing and to check your thyroid function.
* You will complete the questionnaire about kidney cancer care (only during the first 2 years).

Length of Study:

You will take axitinib for up to 12 weeks. You will stop taking axitinib earlier than expected if the disease gets worse or if you have severe side effects. In both cases, you will move on to surgery after axitinib has been stopped.

After surgery, you will be contacted by the study staff every 4 months (+/- 2 weeks) for 1 year, every 6 months (+/- 2 weeks) for the next 2 years and every 12 months (+/- 1 month) for 2 more years (for a total of 5 years after surgery).

This is an investigational study. Axitinib is FDA approved and commercially available to treat advanced kidney cancer in adults when 1 previous drug treatment for this disease has not worked. In this study, it is being used for research purposes.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced renal cell carcinoma without evidence of metastatic disease with absence of adjacent organ invasion or retroperitoneal adenopathy (cT2-T3b, N0, M0). Patients with retroperitoneal lymph nodes </= 2cm in size each are considered N0.
2. Predominant clear cell histology on pre-treatment biopsy of the primary tumor.
3. Patient should be candidate for curative radical nephrectomy.
4. ECOG Performance Status 0-1.
5. Patient must provide signed informed consent.
6. Male or female, age >/= 18 years.
7. Adequate renal function: serum creatinine level </=1.5 x ULN or calculated creatinine clearance (as estimated by GFR using the MDRD formula) is >/= 60 ml/min.
8. Adequate hepatic function: alkaline phosphatase </= 1.5 x ULN; total bilirubin, AST, and ALT </= 1.5 x ULN; INR <1.3 (or <3 if on anticoagulant therapy).
9. Adequate bone marrow function: ANC >/= 1.5 x 10/ 9L; Platelets >/= 100 x 109/L; Hb >9 g/dL
10. Urinary protein <100 on urinalysis (equivalent to <2+ by urine dipstick). If urinalysis protein >/=100 (equivalent to dipstick is >/=2+) then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours
11. No hormonal therapy, chemotherapy, immunotherapy, or any other systemic therapy for a malignancy, in the 5 years prior to current study enrollment.
12. Women of childbearing potential (defined as a female subject who is not surgically sterilized, not at least 1 year postmenopausal) must have negative urine or serum pregnancy test within 4 weeks of enrollment and again on the day of starting therapy and she and/or her partner must utilize birth control while on therapy.
13. Male (defined as a male subject who has not been surgically sterilized) or female patients of child-producing potential must agree to use adequate contraception (e.g. IUD, condom plus spermicide, diaphragm, or cervical cap plus spermicide) or medical contraception: as of date of study enrollment and for at least 1 month after last dose of axitinib. Subjects who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study.

Exclusion Criteria:

1. Evidence of metastatic disease, adjacent organ invasion, retroperitoneal adenopathy on pre-treatment imaging. In addition, patients with inferior vena cava thrombi extending to the atrium or with evidence of Budd-Chiari Syndrome (hepatic dysfunction) will not be eligible for the protocol.
2. Patients who undergo embolization of their primary tumor.
3. Previous treatment for their primary renal tumor, including prior chemotherapy, immunotherapy, targeted therapy, radiation therapy, cryotherapy, radiofrequency ablation or embolization.
4. Active malignancies other than renal cell carcinoma and/or history of other malignancy within the last 5 years, except for adequately treated cone-biopsied in situ carcinoma of the cervix or basal or squamous cell carcinoma of the skin
5. Uncontrolled hypertension (BP>140/90 on medications), as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be </=140 mm Hg, and the baseline diastolic blood pressure readings must be </=90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
6. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, nefazodone, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine).
7. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 or CYP1A2 inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
8. Active gastrointestinal bleeding.
9. Malabsorption syndromes such as celiac disease, cystic fibrosis, inflammatory bowel disease, systemic sclerosis, and carcinoid syndrome.
10. Known HIV or Hepatitis C status.
11. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devise or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
12. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
13. A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
14. Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism
15. Withdrawal of consent.
16. Unwillingness or inability to comply with mandated pretreatment biopsy or therapeutic regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Karam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Karam JA, Devine CE, Urbauer DL, Lozano M, Maity T, Ahrar K, Tamboli P, Tannir NM, Wood CG. Phase 2 trial of neoadjuvant axitinib in patients with locally advanced nonmetastatic clear cell renal cell carcinoma. Eur Urol. 2014 Nov;66(5):874-80. doi: 10.1016/j.eururo.2014.01.035. Epub 2014 Feb 7. PMID 24560330
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 participants consented, but 14 not treated (11 not meeting criteria and 3 declined). Only 25 underwent treatment
Groups:
- Axitinib: 5 mg by mouth twice each day for 12 weeks.
Period: Overall Study
Arm/Group | Axitinib
Started | 25
Completed | 24
Not Completed | 1
Not completed — Non-Compliant with treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 60 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is defined as Complete Response (CR)+ Partial Response (PR) and evaluated when CT abdomen is done after 12 weeks of treatment. Per Response Evaluation Criteria in Solid Tumors Criteria ( RECIST v1.0) Complete Response (CR) is complete disappearance of renal mass; and, Partial Response (PR) is >= 30% decrease in the largest diameter (LD) of the renal mass taking as reference the baseline largest diameter.
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 24
percentage of participants | 28.3 [5.3 to 42.9]

2. Secondary Outcome: Recurrence Free Survival
Description: We will evaluate recurrence-free survival by plotting Kaplan-Meier curves and estimating median recurrence-free survival. RFS is the time from reatment start until death, recurrence or progressive disease, whichever comes first.
Time Frame: After completion of treatment, patients followed w/evaluations every 4 months for 1st year, then every 6 months for next 2 years, yearly until disease progression identified or start of new treatment & yearly survival thereafter until study completion
Population: Anyone who received study treatment
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Axitinib: Participants received 12 weeks of neoadjuvant followed by radical nephrectomy
Arm/Group | Axitinib
Number analyzed (Participants) | 24
Months | 103.1 [49.5 to NA] — Not estimable for the upper found of the 95% Confidence Interval due to insufficient number of participants with events

3. Secondary Outcome: Overall Survival
Description: We will evaluate overall survival by plotting Kaplan-Meier curves and estimating median overall survival. OS is the time from treatment start until death.
Time Frame: From date of randomization until the date of death from any cause, or date of last follow-up, whichever came first, assessed up to 5 years
Population: Anyone who received study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Axitinib: Participants received 12 weeks of neoadjuvant treatment followed by radical nephrectomy
Arm/Group | Axitinib
Number analyzed (Participants) | 24
months | NA [NA to NA] — Not reached for meeting OS and not estimable for the 95% Confidence Interval due to insufficient number of participants with events

4. Secondary Outcome: Postoperative Complications-Any Grade
Description: We used Clavien-Dindo score to record postoperative complications of any grade (Grade 1 thru 5)
Time Frame: From surgery until 30 days after surgery
Population: Anyone who received study treatment and completed the 30-day post-op FU visit
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 23
Participants | 9

5. Secondary Outcome: Surgery-related Complications - High Grade
Description: We used Clavien-Dindo score to record postoperative complications of high grade (Grade 3-5)
Time Frame: From surgery until 30 days after surgery
Population: Anyone who received study treatment and completed the 30-day post-op FU visit
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 23
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 12 weeks. All-Cause Mortality monitored/assessed up to 5 years
Description: No participant deaths reported throughout study.
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 19/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=24)
Hypertension (Vascular disorders) | 19
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 19
Fatigue (General disorders) | 18
Oral mucositis (Gastrointestinal disorders) | 17
Hypothyroidism (Immune system disorders) | 15
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 15
Nausea (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 9
AST/ALT increase (Investigations) | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 4
Myalgias (Immune system disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Gastroesophageal reflux (Gastrointestinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Scrotal skin rash (Skin and subcutaneous tissue disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT01263769/Prot_SAP_000.pdf